CLINICAL TRIAL: NCT04237415
Title: The Effect of Electromyographic (EMG) Biofeedback Training on Electrical Muscle Activity and Functional Status in Zone I-III Flexor Tendon Injuries
Brief Title: Electromyographic (EMG) Biofeedback Training in Zone I-III Flexor Tendon Injuries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, UMUT ERASLAN, Research Assistant, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 60116787-020/50298
Record Dates: First submitted 2020-01-15; First posted 2020-01-23 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Flexor Tendon Rupture; Hand Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMG biofeedback group (Experimental)
  Interventions: Procedure: EMG biofeedback training
- control group (No Intervention)

INTERVENTIONS:
Procedure: EMG biofeedback training
  Arms: EMG biofeedback group

SUMMARY:
Aim: The aim of the study was to investigate the effect of electromyographic (EMG) biofeedback training applied in addition to early passive motion protocol on electrical muscle activity (EMA) and functional status in zone I-III flexor tendon injuries.

Materials and Methods: Cases who underwent surgery for flexor tendon injuries in zone I-III were included in this prospective randomized controlled trial. Cases were randomly divided into two groups of 11 cases each by block randomization. In the first group, EMG biofeedback training was applied in addition to the early passive motion method (modified Duran protocol), while the second group was followed only by early passive motion method. The treatment program was performed by the same physiotherapist three times a week, for 12 weeks. At the postoperative 5th, 12th and 24th weeks, joint range of motion (ROM) and EMA were evaluated, and the Michigan Hand Outcome Questionnaire (MHQ) was administered to the patients. The grip strength at 12th and 24th weeks were also assessed. The Mann-Whitney U Test was used to compare the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Being olunteer,
* No history of neurological, orthopedic, rheumatologic disease or trauma in the related extremity,
* No history of neuropathy due to a metabolic disease (diabetes, etc.),
* Incision of at least one of the FDS or FDP tendons,
* At least one of the FDS or FDP tendons repaired within 2 weeks after the injury,
* No communication problems.

Exclusion Criteria:

* <18 years of age,
* Pregnancy,
* Thumb flexor tendon cuts,
* Digital nerve injury,
* Accompanying fracture, joint capsule injury or skin loss,
* Crush injury,
* Patients with pacemakers,
* Patients with cardiac arrhythmias,
* Epilepsy.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2016-10-10 (Actual); Primary Completion 2018-12-10 (Actual); Study Completion 2019-03-21 (Actual)

PRIMARY OUTCOMES:
Finger joint range of motion | 5th week
  Finger motion was measured by goniometer.Total active motion protocol was used.
Finger joint range of motion | 12th week
  Finger motion was measured by goniometer.Total active motion protocol was used.
Finger joint range of motion | 24th week
  Finger motion was measured by goniometer.Total active motion protocol was used.
Electrical muscle activity | 5th week
  Flexor muscle electrical activity was measured by EMG biofeedback device. For this purpose, surface electrodes were used.
Electrical muscle activity | 12th week
  Flexor muscle electrical activity was measured by EMG biofeedback device. For this purpose, surface electrodes were used.
Electrical muscle activity | 24th week
  Flexor muscle electrical activity was measured by EMG biofeedback device. For this purpose, surface electrodes were used.
Grip strength | 12th week
  Gross and pinch strength were evaluated by hand dynamometer.
Grip strength | 24th week
  Gross and pinch strength were evaluated by hand dynamometer.
Michigan Hand Questionnaire | 5th week
  This questionnaire evaluates the functionality of the hand and consists of 63 questions in total. Each question is scored between 1-5 and the score of each section varies between 0-100. High total score indicates high satisfaction.
Michigan Hand Questionnaire | 12th week
  This questionnaire evaluates the functionality of the hand and consists of 63 questions in total. Each question is scored between 1-5 and the score of each section varies between 0-100. High total score indicates high satisfaction.
Michigan Hand Questionnaire | 24th week
  This questionnaire evaluates the functionality of the hand and consists of 63 questions in total. Each question is scored between 1-5 and the score of each section varies between 0-100. High total score indicates high satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Kitis, PhD, Study Director — Pamukkale University

IPD SHARING:
Plan to Share IPD: No